CLINICAL TRIAL: NCT01100957
Title: Evaluation and Comparison of the New Single Use Ambu aScope With Olympus BF 160 Multiple Use Scope for Securing the Airway of the Anaesthetised/Awake Patients' Normal or Difficult Airway
Brief Title: Evaluation of the Single Use Flexible Optical Scope Versus Multiple Use Flexible Optical Scopes for Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Michael Seltz Kristensen, M.D., Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: aScope-1+2 a; H-A-2009-022
Record Dates: First submitted 2010-03-25; First posted 2010-04-09 (Estimated); Last update posted 2011-08-24 (Estimated); Status verified 2010-03

CONDITIONS: Tracheal Intubation; Difficult Airway
MeSH Terms: interventions — Intubation, Intratracheal

ARMS (2):
- Conventional flexible videoscope for intubation (Active Comparator)
  Interventions: Procedure: tracheal intubation with a single use flexible videoscope
- Single-patient flexible endoscope (Experimental): Single-patient flexible video-endoscope used for tracheal intubation in this intervention-arm
  Interventions: Procedure: tracheal intubation with a single use flexible videoscope

INTERVENTIONS:
Procedure: tracheal intubation with a single use flexible videoscope — tracheal intubation with a single use flexible videoscope

SUMMARY:
The study is in two parts

Part one of the study describes the use of the new single-use flexible video-scope for intubation of patients with predicted normal airways.

Part two compares the performance of the single-use flexible video-scope with that of a conventional flexible video-scope for awake intubation of patients with predicted difficult airways.

The hypothesis is that the new single-use flexible video-scope for intubation performs as well as the traditional scope.

ELIGIBILITY:
Inclusion Criteria:

1. Study part 1:

   * Patients scheduled for tracheal intubation and predicted to have a normal airway
   * ASA class I, II or III
   * >18 years
2. Study part 2:

   * Adult patients scheduled for tracheal intubation and predicted to have a difficult airway
   * ASA class I, II or III
   * >18 years

Exclusion Criteria:

1. Study part 1:

   * Massive bleeding from the mouth
   * Previously abandoned flexible optical intubation
2. Study part 2:

   * Massive bleeding from the mouth
   * Previously abandoned flexible optical intubation
   * Patients with audible stridor
   * Patients with dyspnea

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
time for completion of intubation | September 2010
  This, the time for intubation, is measured immediately during the intubation, on the day that the specific patient participates in the study

SECONDARY OUTCOMES:
time for preparing and cleaning the endoscopes | september 2010
  this is measured in the hour before and after the intubation
number of intubation attempts | september 2010
  measured during the intubation
success rate of endotracheal intubation | september 2010
  measured during the intubation
total time for the intubation-procedure inclusive the time for distributing local analgesics | september 2010
  measured during the intubation
Quality of the image from the videoscope | september 2010
  Observed immediately before, and during, the intubation
Evaluation of the insertion cord of the flexible scope | september 2010
  measured during the intubation
Evaluation of the working-/-injection-channel | september 2010
  measured during the intubation

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Kristensen, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, section for anaesthesia for ENT and Maxillofacial surgery, section 3071, Copenhagen, Denmark